CLINICAL TRIAL: NCT01737957
Title: Safety and Efficacy of Single-session, Low-fluence Panretinal Photocoagulation (PRP) for Proliferative Diabetic Retinopathy (PDR)
Brief Title: Safety and Efficacy of Low-Fluence PRP for PDR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: APEC-LFPRP
Record Dates: First submitted 2012-11-23; First posted 2012-11-30 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic retinopathy; Pan-retinal photocoagulation
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-fluence (Experimental): Low-fluence pan-retinal photocoagulation in a single session for proliferative diabetic retinopathy
  Interventions: Device: Low-fluence PRP with 532nm green LASER
- Full-fluence (Active Comparator): Full-fluence pan-retinal photocoagulation for proliferative diabetic retinopathy
  Interventions: Device: Full-Fluence PRP with 532nm LASER

INTERVENTIONS:
Device: Low-fluence PRP with 532nm green LASER — To administer low-fluence PRP in a single session for PDR
  Other Names: PURE-POINT LASER
  Arms: Low-fluence
Device: Full-Fluence PRP with 532nm LASER — To administer full-fluence PRP in two sessions for PDR
  Other Names: PURE-POINT LASER
  Arms: Full-fluence

SUMMARY:
To determine the safety and efficacy of a single session of low-fluence panretinal photocoagulation when compared to full-fluence PRP. Hypothesis: a single-session of low-fluence PRP will be safe regarding the progression of macular edema and the presence of adverse events, and will efficiently induce regression of neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetics
* Proliferative diabetic retinopathy

Exclusion Criteria:

* Previous treatment with PRP
* Media opacities
* Previous treatment for macular edema (LASER or intravitreal injections)
* Recent (less than 6 months) ophthalmic surgery
* Only eyes
* Intra-retinal or sub-retinal fluid with foveal involvement
* Chronic renal failure
* History of liver or pancreatic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Macular thickness change | Base-line, 1 week, 6 weeks, 12 weeks, 16 weeks
  Measurement of macular thickness changes by spectral domain optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Adverse events | 16 weeks
  Presence or absence of adverse events

OTHER OUTCOMES:
Regression of neovessels, change over time | Base-line, 1 week, 6 weeks, 12 weeks, 16 weeks
  Regression of neovessels observed by fluorescein angiography

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Salcedo-Villanueva, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación Para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico